CLINICAL TRIAL: NCT04848532
Title: Does Aberrant Decision Making Prevent Success in Adolescent Behavioral Weight Loss Treatment?
Brief Title: Problematic Decision-Making and Adolescent Weight Loss
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2005007834
Record Dates: First submitted 2021-03-17; First posted 2021-04-19 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Overweight Adolescents; Overweight or Obesity; Impulsive Behavior; Overeating
MeSH Terms: conditions — Overweight; Obesity; Impulsive Behavior; Hyperphagia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adolescent-specific behavioral weight loss treatment (Experimental)
  Interventions: Behavioral: Weight loss treatment

INTERVENTIONS:
Behavioral: Weight loss treatment — The intervention will consist of group-based, weekly or biweekly weight loss coaching (75 minutes per session), which will occur via Zoom videoconferencing software. This intervention is designed to facilitate a 5-10% weight loss and engagement in up to 250 min/week of moderate-to-vigorous physical activity, which is the standard recommendation in lifestyle modification programs for adolescents. Participants will also be asked to download and utilize the smartphone app, Fitbit, to track eating behavior. Weight loss coaches will be experts in lifestyle modification who have graduate degrees in psychology or a related field. Participants will be given guidance on how to reduce your calorie intake (using a balanced deficit diet) and gradually increase your physical activity. Participants will learn to set goals for diet, weight, and physical activity.
  Other Names: Lifestyle modification

SUMMARY:
This study evaluates the associations between baseline decision-making processes, engagement in problematic dietary practices, and post-intervention weight loss outcomes among adolescents. Results from the study will provide specific direction for what components should comprise future decision-making interventions for adolescents with overweight/obesity.

DETAILED DESCRIPTION:
Adolescent overweight and obesity (AOB; i.e., a body mass index (BMI) greater than 85th percentile for age, height, and gender) affects 34.5% of adolescents. Over 80% of obese adolescents will become obese adults and experience increased risk of cardiovascular disease, type 2 diabetes, gallbladder disease, and some forms of cancer. Because of contraindications and hesitations to pursue psychopharmacology or bariatric surgery, behavioral interventions are the first-line treatment for AOB. Unfortunately, adolescent outcomes from pediatric behavioral obesity treatments are poor. In fact, the modal weight loss in behavioral interventions is less than a single BMI point, and many participants lose no weight at all. Outcomes in adolescents are worse than those found in younger children and adults. Notably, the vast majority of existing interventions tested in adolescents are designed for younger children, which may preclude an adolescent's success in these interventions. Successful behavioral AOB interventions may require augmentations that address developmental concerns unique to adolescence. For example, research has shown that, in contrast to younger children, many adolescents are making their own food decisions and are thus more likely to engage in problematic eating behaviors during treatment. As a necessary step towards developing specialized interventions for AOB, it is critical to understand the underlying mechanisms of continued engagement in problematic eating behaviors during AOB interventions.

Three types of problematic eating behaviors are strongly linked (cross-sectionally and longitudinally) with AOB. First, reward-driven overeating (i.e., frequently eating energy-dense foods) results in excess calorie intake, which, in turn, produces adiposity during childhood and adolescence. Second, loss-of-control eating (LOC; the experience of not being able to stop eating once started) is an exceptionally strong predictor of excess weight gain, i.e., an additional 2.4kg per year compared to peers without LOC. Third, rigid dietary restriction involves skipping meals and cutting out food groups for the purposes of weight regulation, but instead results in intense feelings of deprivation. As a result, rigid dietary restriction has the paradoxical effect of calorie overconsumption, excess weight gain, and poor outcomes from pediatric obesity treatment. Taken together, findings indicate that elucidating the drivers of these three problematic eating behaviors is critical to improving AOB treatment outcomes.

An aberrant decision-making framework represents an attractive paradigm for understanding the above-described problematic eating behaviors, especially given that they all run counter to adolescents' intentions and well-being. There are several aberrant decision-making processes endemic to the adolescent developmental period. Three of these processes in particular appear to be directly linked to the three problematic eating behaviors described above. To the extent that aberrant decision-making produces problematic eating behavior, aberrant decision-making can also be hypothesized to predict poor weight loss outcomes. Below, three aberrant decision-making processes and their links to problematic eating behavior are described.

Increased delay discounting. Delay discounting refers to the tendency to discount greater, later rewards in favor of smaller, sooner rewards. A combination of greater sensitivity to reward and slow development of self-regulatory neural processes contributes to especially high discounting rates in some adolescents. Relatively higher discounting rates may produce reward-driven eating, i.e., frequent consumption of energy-dense foods (e.g., high-fat, high sugar foods), while discounting the future reward (e.g., weight loss) that would be derived from forgoing immediate gratification. Indeed, a recent meta-analysis concluded that higher discounting rates were strongly cross-sectionally linked with AOB. Although behavioral weight loss programs discourage consumption of energy-dense foods, psychological strategies for how to prioritize long-term over short-term rewards are not provided. Thus, delay discounting likely contributes to continued reward-driven eating during treatment. However, no studies have tested whether delay discounting predicts reward-driven overeating (and its effect on weight) during AOB treatment.

Affect-driven impulsivity. Affect-driven impulsivity refers to a tendency to choose maladaptive behaviors geared towards the immediate cessation of a negative affective state, despite negative consequences. Affect-driven impulsivity likely drives continued LOC eating during treatment, precluding successful weight loss. Affect-driven impulsivity is a cross-sectional predictor of AOB, but it may be a particularly strong driver of LOC eating because compulsive eating serves the function of reducing distress. Although no studies have compared adolescents with and without LOC on affect-driven impulsivity, adolescents with LOC eating demonstrate overall higher levels of emotional reactivity and emotional eating. LOC eating resulting from affect-driven impulsivity may continue to occur during treatment because little treatment content focuses on skills for tolerating negative affect. Dr. Manasse's work demonstrates that increased affect-driven impulsivity predicts poor outcomes from adult binge eating treatment. However, no studies have examined whether affect-driven impulsivity predicts (1) engagement in LOC during treatment or (2) poor AOB treatment outcomes.

Perseverative decision-making. Perseverative decision-making is characterized by weakened ability to stop engagement in habitual behaviors despite changing contingencies. Highly perseverative decision-making may contribute to repeated engagement in rigid dietary restriction (i.e., setting rigid calorie goals, cutting out specific foods) that increase deprivation. This deprivation, in turn, leads to episodes of overeating that preclude successful caloric restriction. Those who show highly perseverative decision-making continue engaging in this rigid dietary restriction behavior despite the fact that it ultimately delivers the opposite of its intended effect. Indeed, perseverative decision-making and rigid dieting are associated with the presence of LOC eating, and perseveration is cross-sectionally associated with obesity in adolescence. Despite the established links between perseverative decision-making with unhealthy dieting and excess weight, no studies have examined whether perseverative decision-making underlies continued engagement in problematic dietary restriction during treatment and predicts poor outcomes.

To inform the development of tailored intervention approaches, the current study, funded by the National Institutes of Health, aims to elucidate the specific aberrant decision-making processes associated with three problematic eating behaviors and weight loss outcomes. Results from the study will provide specific direction for what components (e.g., strategies for tolerating emotional distress or promoting flexible thinking) should comprise a future decision-making intervention for AOB and for whom (e.g., those with LOC, those who engage in problematic restriction) certain components would be most relevant. Given that LOC eating is a robust predictor of excess weight gain but only 20-30% of those with AOB endorse LOC eating, the study team will oversample individuals with clinically significant LOC, i.e., the study will recruit a total of 80 adolescents (ages 14-18) with overweight/obesity, half of whom (n=40) endorse clinically significant (i.e., at least once weekly) LOC eating and the other half of whom (n=40) endorse subclinical LOC or no LOC. All participants will receive a 16-week group-based, remotely delivered behavioral weight loss intervention and complete a 6-month follow-up. Decision-making measures will be administered at baseline. Problematic eating behaviors and weight will be assessed at all time points.

ELIGIBILITY:
Inclusion Criteria:

1. Are between 14 and 18 years of age
2. Have a BMI between the 85th and 99th percentiles for sex and age as determined by the CDC growth charts
3. Are currently living at home with a parent or guardian
4. Have at least one parent or guardian who is willing to participate in the study
5. Are willing to complete baseline assessment tasks
6. Have a smartphone, are willing to download an app to track food intake and complete surveys on the phone for two seven-day periods throughout the course of the study, and are willing to wear a fitness tracker during these same two week-long periods
7. Are located in the US and wiling/able to participate in remote intervention and assessments

Exclusion Criteria:

1. Acute suicide risk
2. Inability to engage in physical activity (defined as walking two city blocks without stopping)
3. Have diabetes or a history of bariatric surgery
4. Current medical or psychiatric condition that may pose a risk to the participant during intervention, cause a change in weight, or limit ability to comply with the program (i.e., bulimia nervosa, substance abuse disorder, psychosis, bipolar I disorder, and/or any condition prohibiting physical activity)
5. Are pregnant or planning to become pregnant in the next 2 years
6. Recently began or changed the dose of a medication that can cause significant change in weight
7. Have experienced weight loss ≥ 5% in the previous 6 months
8. Are planning to begin in the next 16 months, or are currently participating in, another weight loss treatment or psychotherapy for binge eating and/or weight loss
9. Are engaging in compensatory vomiting, other severe compensatory behaviors, or more than 12 of any compensatory behaviors in the previous 3 months
10. Are currently taking medication (e.g., Contrave, Alli, etc.) which is specifically intended for weight loss

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Percent of 95 percentile BMI | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Manasse, Ph.D., Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-26): https://cdn.clinicaltrials.gov/large-docs/32/NCT04848532/Prot_SAP_000.pdf